CLINICAL TRIAL: NCT00460811
Title: A Randomized, Multicenter, Double-blind, Placebo-controlled, Dose-range-finding, Parallel-design, Phase 2 Trial of Oral Linaclotide Acetate Administered to Patients With Irritable Bowel Syndrome With Constipation
Brief Title: Randomized, Double-blind, Dose-range-finding, Phase 2 Study of Linaclotide Administered to Patients With Irritable Bowel Syndrome With Constipation (IBS-C)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCP-103-202
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Irritable Bowel Syndrome With Constipation
Keywords: Irritable Bowel Syndrome with Constipation; IBS; Irritable Bowel Syndrome; linaclotide acetate; linaclotide; MD-1100
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- 72 ug linaclotide acetate (Active Comparator)
  Interventions: Drug: Linaclotide Acetate
- 145 ug linaclotide acetate (Active Comparator)
  Interventions: Drug: Linaclotide Acetate
- 290 ug linaclotide acetate (Active Comparator)
  Interventions: Drug: Linaclotide Acetate
- 579 ug linaclotide acetate (Active Comparator)
  Interventions: Drug: Linaclotide Acetate
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Linaclotide Acetate — Oral, once daily
  Arms: 145 ug linaclotide acetate; 290 ug linaclotide acetate; 579 ug linaclotide acetate; 72 ug linaclotide acetate
Drug: Matching placebo — Oral, once daily
  Arms: Matching Placebo

SUMMARY:
The purpose of this study is to determine the safety, efficacy, and dose response of a range of oral doses of linaclotide administered to patients meeting criteria for IBS-C.

ELIGIBILITY:
Inclusion Criteria:

* Must not be pregnant or breastfeeding and agree to use birth control;
* Completion of a negative colonoscopy as per American Gastroenterology Association (AGA) criteria and no clinically-significant laboratory or physical examination findings;
* Meets protocol-defined criteria for IBS-C, including stool frequency, straining, stool consistency, abdominal pain, and abdominal discomfort criteria;
* Demonstrates English fluency and has access to a touch-tone telephone.

Exclusion Criteria:

* Recent history of mushy or watery stools;
* Various medical conditions, medical histories, or family medical histories that would not make the patient a good candidate for the study;
* Clinically-significant alarm symptoms;
* Secondary causes of constipation or evacuation disorders;
* Surgery to the gastrointestinal tract;
* Usage of prohibited medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2007-04; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Microbia Medical Director, MD, Study Director — Microbia, Inc.
Locations (85):
- United States (79):
  - Microbia Investigational Site, Huntsville, Alabama
  - Microbia Investigational Site, Chandler, Arizona
  - Microbia Investigational Site, Tuscon, Arizona
  - Microbia Investigational Site, Sherwood, Arkansas
  - Microbia Investigational Site, Anaheim, California
  - Microbia Investigational Site, Garden Grove, California
  - Microbia Investigational Site, Sacramento, California
  - Microbia Investigational Site, San Diego, California
  - Microbia Investigational Site, Bristol, Connecticut
  - Microbia Investigational Site, Boynton Beach, Florida
  - Microbia Investigational Site, Dunedin, Florida
  - Microbia Investigational Site, Largo, Florida
  - Microbia Investigational Site, Ocala, Florida
  - Microbia Investigational Site, Port Orange, Florida
  - Microbia Investigational Site, Stuart, Florida
  - Microbia Investigational Site, Tampa, Florida
  - Microbia Investigational Site, Stockbridge, Georgia
  - Microbia Investigational Site, Libertyville, Illinois
  - Microbia Investigational Site, Peoria, Illinois
  - Microbia Investigational Site, Clive, Iowa
  - Microbia Investigational Site, Davenport, Iowa
  - Microbia Investigational Site, Mission, Kansas
  - Microbia Investigational Site, Shawnee, Kansas
  - Microbia Investigational Site, Baton Rouge, Louisiana
  - Microbia Investigational Site, Monroe, Louisiana
  - Microbia Investigational Site, West Monroe, Louisiana
  - Microbia Investigational Site, Annapolis, Maryland
  - Microbia Investigational Site, Silver Spring, Maryland
  - Microbia Investigational Site, Fall River, Massachusetts
  - Microbia Investigational Site, Ann Arbor, Michigan
  - Microbia Investigational Site, St Louis, Missouri
  - Microbia Investigational Site, Missoula, Montana
  - Microbia Investigational Site, Henderson, Nevada
  - Microbia Investigational Site, Las Vegas, Nevada
  - Microbia Investigational Site, Blackwood, New Jersey
  - Microbia Investigational Site, Great Neck, New York
  - Microbia Investigational Site, Pittsford, New York
  - Microbia Investigational Site, Asheville, North Carolina
  - Microbia Investigational Site, Chapel Hill, North Carolina
  - Microbia Investigational Site, Elkin, North Carolina
  - Microbia Investigational Site, Greensboro, North Carolina
  - Microbia Investigational Site, Harrisburg, North Carolina
  - Microbia Investigational Site, Hickory, North Carolina
  - Microbia Investigational Site, Raleigh, North Carolina
  - Microbia Investigational Site, Statesville, North Carolina
  - Microbia Investigational Site, Winston-Salem, North Carolina
  - Microbia Investigational Site, Cincinnati, Ohio
  - Microbia Investigational Site, Cleveland, Ohio
  - Microbia Investigational Site, Dayton, Ohio
  - Microbia Investigational Site, Sylvania, Ohio
  - Microbia Investigational Site, Oklahoma City, Oklahoma
  - Microbia Investigational Site, Tulsa, Oklahoma
  - Microbia Investigational Site, Yukon, Oklahoma
  - Microbia Investigational Site, Medford, Oregon
  - Microbia Investigational Site, Levittown, Pennsylvania
  - Microbia Investigational Site, Pittsburgh, Pennsylvania
  - Microbia Investigational Site, Reading, Pennsylvania
  - Microbia Investigational Site, Sellersville, Pennsylvania
  - Microbia Investigational Site, Anderson, South Carolina
  - Microbia Investigational Site, Mt. Pleasant, South Carolina
  - Microbia Investigational Site, Simpsonville, South Carolina
  - Microbia Investigational Site, Summerville, South Carolina
  - Microbia Investigational Site, Bristol, Tennessee
  - Microbia Investigational Site, Germantown, Tennessee
  - Microbia Investigational Site, Jackson, Tennessee
  - Microbia Investigational Site, Kingsport, Tennessee
  - Microbia Investigational Site, Beaumont, Texas
  - Microbia Investigational Site, Corsicana, Texas
  - Microbia Investigational Site, El Paso, Texas
  - Microbia Investigational Site, San Antonio, Texas
  - Microbia Investigational Site, Ogden, Utah
  - Microbia Investigational Site, Chesapeake, Virginia
  - Microbia Investigational Site, Lynchburg, Virginia
  - Microbia Investigational Site, Richmond, Virginia
  - Microbia Investigational Site, Lakewood, Washington
  - Microbia Investigational Site, Olympia, Washington
  - Microbia Investigational Site, Vancouver, Washington
  - Microbia Investigational Site, Charleston, West Virginia
  - Microbia Investigational Site, La Crosse, Wisconsin
- Canada (6):
  - Microbia Investigational Site, Abbortsford, British Columbia
  - Microbia Investigational Site, Winnipeg, Manitoba
  - Microbia Investigational Site, Guelph, Ontario
  - Microbia Investigational Site, Milton, Ontario
  - Microbia Investigational Site, Toronto, Ontario
  - Microbia Investigational Site, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Lembo A, Kuo B, Boinpally R, Li E, Mallick M, Bochenek W, Bartolini W. Randomised clinical trial: effects of MD-7246 on irritable bowel syndrome with diarrhoea. Aliment Pharmacol Ther. 2023 Jan;57(2):192-204. doi: 10.1111/apt.17274. Epub 2022 Nov 2. PMID 36324245
- [Derived] Johnston JM, Kurtz CB, Macdougall JE, Lavins BJ, Currie MG, Fitch DA, O'Dea C, Baird M, Lembo AJ. Linaclotide improves abdominal pain and bowel habits in a phase IIb study of patients with irritable bowel syndrome with constipation. Gastroenterology. 2010 Dec;139(6):1877-1886.e2. doi: 10.1053/j.gastro.2010.08.041. Epub 2010 Aug 27. PMID 20801122

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred over a 12 month period from March 2007 to February 2008 at 92 US study sites.
Pre-assignment Details: Patients went through a 14 to 17 day Pretreatment Period during which the patients provided qualifying bowel habit and symptoms, and rescue medicine usage information through an interactive voice response system (IVRS).
Groups:
- 72 μg Linaclotide Acetate: Linaclotide, 72μg dose, oral administration, once per day
- 145 μg Linaclotide Acetate: Linaclotide, 145μg dose, oral administration, once per day
- 290 μg Linaclotide Acetate: Linaclotide, 290μg dose, oral administration, once per day
- 579 μg Linaclotide Acetate: Linaclotide, 579μg dose, oral administration, once per day
- Matching Placebo: Dose-matched placebo, oral administration, once per day
Period: Overall Study
Arm/Group | 72 μg Linaclotide Acetate | 145 μg Linaclotide Acetate | 290 μg Linaclotide Acetate | 579 μg Linaclotide Acetate | Matching Placebo
Started | 79 | 82 | 85 | 89 | 85
Completed | 63 | 67 | 71 | 71 | 65
Not Completed | 16 | 15 | 14 | 18 | 20
Not completed — Adverse Event | 4 | 6 | 3 | 10 | 2
Not completed — Noncompliance | 1 | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 7 | 7 | 6 | 3 | 11
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 5 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- 72 µg Linaclotide Acetate: Linaclotide, 72μg dose, oral administration, once per day
- 145 µg Linaclotide Acetate: Linaclotide, 145μg dose, oral administration, once per day
- 290 µg Linaclotide Acetate: Linaclotide, 290μg dose, oral administration, once per day
- 579 µg Linaclotide Acetate: Linaclotide, 579μg dose, oral administration, once per day
- Total: Total of all reporting groups
Arm/Group | 72 µg Linaclotide Acetate | 145 µg Linaclotide Acetate | 290 µg Linaclotide Acetate | 579 µg Linaclotide Acetate | Matching Placebo | Total
Number analyzed (Participants) | 79 | 82 | 85 | 89 | 85 | 420
Age Continuous [Mean (Standard Deviation); unit: years] | 42.3 (12.5) | 45.6 (10.8) | 45.8 (11.4) | 43.7 (11.4) | 44.3 (11.3) | 44.4 (11.5)
Age, Customized [Number; unit: Participants]
  18 years to 65 years | 77 | 79 | 81 | 86 | 85 | 408
  Older than 65 years | 2 | 3 | 4 | 3 | 0 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 78 | 78 | 79 | 78 | 387
  Male | 5 | 4 | 7 | 10 | 7 | 33
Region of Enrollment [Number; unit: participants]
  United States | 75 | 79 | 80 | 86 | 81 | 401
  Canada | 4 | 3 | 5 | 3 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly Normalized Complete Spontaneous Bowel Movement (CSBM) Rate During Weeks 1 Through 12 of the Treatment Period
Description: The change in the weekly normalized CSBM Rate during Weeks 1 through 12 of the Treatment Period from the weekly normalized CSBM Rate obtained during the Pretreatment Period.
  The CSBM rate was normalized based on the number of CSBMs occurring in that week, adjusting for differences in the duration of the week and black-out periods (time not covered due to a missed IVRS call) versus 7x24 hours.
Time Frame: Change from Baseline to Week 12
Population: The Intent-to-treat (ITT) Population included 419 patients of the Safety Population who also had ≥ 1 post-dose evaluation of the primary efficacy assessment (i.e., CSBM Frequency)
Measure: Least Squares Mean (Standard Error); unit: CSBMs per week
Groups:
- 72 ug Linaclotide Acetate: Linaclotide, 72μg dose, oral administration, once per day
- 145 ug Linaclotide Acetate: Linaclotide, 145μg dose, oral administration, once per day
- 290 ug Linaclotide Acetate: Linaclotide, 290μg dose, oral administration, once per day
- 579 ug Linaclotide Acetate: Linaclotide, 579μg dose, oral administration, once per day
Arm/Group | 72 ug Linaclotide Acetate | 145 ug Linaclotide Acetate | 290 ug Linaclotide Acetate | 579 ug Linaclotide Acetate | Matching Placebo
Number analyzed (Participants) | 79 | 82 | 84 | 89 | 85
CSBMs per week | 2.90 (0.385) | 2.49 (0.380) | 3.61 (0.372) | 2.68 (0.369) | 1.01 (0.372)
Statistical Analysis 1: Comparison: 72 ug Linaclotide Acetate vs Matching Placebo; For each of the 4 active linaclotide groups, the null hypothesis was that there was no difference between placebo and the dose group in the change from baseline in the weekly normalized CSBM Rate. An observed cases (OC) approach to missing post-baseline data was applied: any missing data were not imputed; Test type: Superiority or Other; p = 0.0002, ANCOVA
Statistical Analysis 2: Comparison: 145 ug Linaclotide Acetate vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0036, ANCOVA
Statistical Analysis 3: Comparison: 290 ug Linaclotide Acetate vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 4: Comparison: 579 ug Linaclotide Acetate vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0008, ANCOVA

2. Secondary Outcome: CSBM 75% Responder for the Treatment Period (Based on the Normalized Rate)
Description: For each week of the Treatment and Posttreatment Periods, a patient was considered a CSBM Responder if for that week the patient 1) completed ≥ 4 days of IVRS questions, 2) had a CSBM rate of ≥ 3 for the week, and 3) had an increase in CSBM rate of ≥ 1 from the baseline weekly CSBM rate.
Time Frame: Change from Baseline to Week 12
Population: The ITT Population included 419 patients of the Safety Population who also had ≥ 1 post-dose evaluation of the primary efficacy assessment (i.e., CSBM Frequency).
Measure: Number; unit: participants
Arm/Group | 72 μg Linaclotide Acetate | 145 μg Linaclotide Acetate | 290 μg Linaclotide Acetate | 579 μg Linaclotide Acetate | Matching Placebo
Number analyzed (Participants) | 79 | 82 | 84 | 89 | 85
participants | 20 | 16 | 27 | 21 | 10

3. Secondary Outcome: Change From Baseline in the Weekly Normalized SBM Rate for the Treatment Period
Description: SBMs were measured daily during the treatment period by patient calls to the IVRS.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: SBMs per week
Arm/Group | 72 ug Linaclotide Acetate | 145 ug Linaclotide Acetate | 290 ug Linaclotide Acetate | 579 ug Linaclotide Acetate | Matching Placebo
Number analyzed (Participants) | 79 | 82 | 84 | 89 | 85
SBMs per week | 4.62 (0.457) | 4.36 (0.453) | 4.97 (0.442) | 5.64 (0.439) | 1.68 (0.442)

4. Secondary Outcome: Change From Baseline in Stool Consistency (7-point Ordinal BSFS) for the Treatment Period
Description: Stool consistency analyses were performed using the 7-point Bristol Stool Form Scale (BSFS), whereby a score of 1 = separate hard lumps like nuts (difficult to pass); 2 = sausage shaped but lumpy; 3 = like a sausage but with cracks on surface; 4 = like a sausage or snake, smooth and soft; 5 = soft blobs with clear-cut edges (passed easily); 6 = fluffy pieces with ragged edges, a mushy stool; and 7 = watery, no solid pieces (entirely liquid).
Time Frame: Change from Baseline to Week 12
Population: The ITT Population included 419 patients of the Safety Population who also had ≥ 1 post-dose evaluation of the primary efficacy assessment (i.e., CSBM Frequency). 15 patients with no pretreatment spontaneous bowel movements were excluded from the Stool Consistency analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 72 μg Linaclotide Acetate | 145 μg Linaclotide Acetate | 290 μg Linaclotide Acetate | 579 μg Linaclotide Acetate | Matching Placebo
Number analyzed (Participants) | 76 | 78 | 82 | 85 | 83
units on a scale | 1.91 (0.133) | 1.80 (0.131) | 2.28 (0.127) | 2.20 (0.127) | 0.56 (0.127)

5. Secondary Outcome: Change From Baseline in Straining (5-point Ordinal Scale) for the Treatment Period
Description: Straining was assessed using a 5-point ordinal scale, whereby a score of 1 = not at all, 2 = a little bit, 3 = a moderate amount, 4 = a great deal, and 5 = an extreme amount.
Time Frame: Change from Baseline to Week 12
Population: The ITT Population included 419 patients of the Safety Population who also had ≥ 1 post-dose evaluation of the primary efficacy assessment (i.e., CSBM Frequency). 15 patients with no pretreatment spontaneous bowel movements were excluded from the Straining analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 72 μg Linaclotide Acetate | 145 μg Linaclotide Acetate | 290 μg Linaclotide Acetate | 579 μg Linaclotide Acetate | Matching Placebo
Number analyzed (Participants) | 76 | 78 | 82 | 85 | 83
units on a scale | -1.23 (0.081) | -1.20 (0.080) | -1.48 (0.077) | -1.35 (0.078) | -0.71 (0.078)

6. Secondary Outcome: Change From Baseline in Degree of Relief of Irritable Bowel Syndrome (IBS) Symptoms (7-point Balanced Scale) for the Treatment Period
Description: Patients provided a weekly assessment of Degree of Relief of IBS Symptoms using a 7-point balanced scale (1=completely relieved, 2=considerably relieved, 3=somewhat relieved, 4=unchanged, 5=somewhat worse, 6=considerably worse, 7=as bad as I can imagine).
Time Frame: Change from Baseline to Week 12
Population: The ITT Population included 419 patients of the Safety Population who also had ≥ 1 post-dose evaluation of the primary efficacy assessment (i.e., CSBM Frequency). 13 patients who dropped out prior to finishing 1 week of the trial have missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 72 μg Linaclotide Acetate | 145 μg Linaclotide Acetate | 290 μg Linaclotide Acetate | 579 μg Linaclotide Acetate | Matching Placebo
Number analyzed (Participants) | 77 | 79 | 81 | 87 | 82
units on a scale | -1.33 (0.108) | -1.37 (0.107) | -1.66 (0.105) | -1.49 (0.104) | -0.81 (0.105)

7. Secondary Outcome: Change From Baseline in Abdominal Pain (5-point Ordinal Scale) for the Treatment Period
Description: During the study, patients provided their self assessment of abdominal pain using a 5-point ordinal scale (1=none, 2=mild, 3=moderate, 4=severe, 5=very severe
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 72 μg Linaclotide Acetate | 145 μg Linaclotide Acetate | 290 μg Linaclotide Acetate | 579 μg Linaclotide Acetate | Matching Placebo
Number analyzed (Participants) | 79 | 82 | 84 | 89 | 85
units on a scale | -0.71 (0.075) | -0.71 (0.074) | -0.90 (0.073) | -0.86 (0.072) | -0.49 (0.073)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from March of 2007 to April 2008.
Arm/Group | 72 µg Linaclotide Acetate | 145 µg Linaclotide Acetate | 290 µg Linaclotide Acetate | 579 µg Linaclotide Acetate | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/82 | 1/85 | 0/89 | 0/85
Other Adverse Events (participants affected / at risk) | 21/79 | 23/82 | 26/85 | 30/89 | 17/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 72 µg Linaclotide Acetate (N=79) | 145 µg Linaclotide Acetate (N=82) | 290 µg Linaclotide Acetate (N=85) | 579 µg Linaclotide Acetate (N=89) | Matching Placebo (N=85)
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 72 µg Linaclotide Acetate (N=79) | 145 µg Linaclotide Acetate (N=82) | 290 µg Linaclotide Acetate (N=85) | 579 µg Linaclotide Acetate (N=89) | Matching Placebo (N=85)
Abdominal distension (Gastrointestinal disorders) | 1 | 3 | 1 | 4 | 5
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 4 | 7 | 3
Diarrhea (Gastrointestinal disorders) | 9 | 10 | 14 | 16 | 1
Headache (Nervous system disorders) | 1 | 3 | 5 | 2 | 6
Nasopharyngitis (Infections and infestations) | 3 | 7 | 1 | 1 | 5
Nausea (Gastrointestinal disorders) | 1 | 8 | 1 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 4 | 5 | 3
Urinary tract infection (Infections and infestations) | 7 | 1 | 5 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that publication cannot be made for 24 months from the date of final data lock of the study, the sponsor can review the publication prior to public release, sponsor requires a minimum 60 day review period for each publication, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request an additional delay period of 60 days in order to protect potentially patentable information.